CLINICAL TRIAL: NCT00230971
Title: A Multicenter, Open-Label, Randomized Comparative Study of Tigecycline vs Ceftriaxone Sodium Plus Metronidazole for the Treatment of Hospitalized Subjects With Complicated Intra-abdominal Infection
Brief Title: Study Comparing Tigecycline Versus Ceftriaxone Sodium Plus Metronidazole in Complicated Intra-abdominal Infection (cIAI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3074A1-315
Record Dates: First submitted 2005-09-30; First posted 2005-10-03 (Estimated); Results first posted 2010-04-26 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Appendicitis; Cholecystitis; Diverticulitis; Intra-Abdominal Abscess; Intra-Abdominal Infection; Peritonitis
Keywords: Intra-Abdominal Infections; Abscess
MeSH Terms: conditions — Appendicitis; Cholecystitis; Diverticulitis; Abdominal Abscess; Intraabdominal Infections; Peritonitis; Abscess | interventions — Tigecycline; Ceftriaxone; Metronidazole

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: tigecycline
- B (Active Comparator)
  Interventions: Drug: ceftriaxone plus metronidazole

INTERVENTIONS:
Drug: tigecycline — every 12 hours IV (an initial dose of 100 mg followed by 50 mg every 12 hours)
  Arms: A
Drug: ceftriaxone plus metronidazole — Ceftriaxone sodium 2 g once daily intravenously plus metronidazole 1 g to 2 g daily given in divided doses intravenously. Test article should be administered for a minimum of 4 days and up to 14 days at the discretion of the investigator.
  Arms: B

SUMMARY:
This is a study of the safety and efficacy of tigecycline to ceftriaxone sodium plus metronidazole in hospitalized subjects with cIAI. Subjects will be followed for efficacy through the test-of-cure assessment. Safety evaluations will occur through the treatment and post-treatment periods and continue through resolution or stability of the adverse event(s).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of complicated intra-abdominal infection that requires surgery within 24 hours.
* Fever plus other symptoms such as nausea, vomiting, abdominal pain.

Exclusion Criteria:

* Cancer
* Medicines that suppress the immune system
* Dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2005-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Australia, China, Hong Kong, medinfo@wyeth.com; Trial Manager, Principal Investigator — For Taiwan, medinfo@wyeth.com; Trial Manager, Principal Investigator — For Denmark, Finland, MedInfoNord@wyeth.com; Trial Manager, Principal Investigator — For Germany, MedinfoDEU@wyeth.com; Trial Manager, Principal Investigator — For South Africa, ZAFinfo@wyeth.com; Trial Manager, Principal Investigator — For Italy, Greece, decresg@wyeth.com; Trial Manager, Principal Investigator — For UK, ukmedinfo@wyeth.com; Trial Manager, Principal Investigator — For Switzerland, med@wyeth.com; Trial Manager, Principal Investigator — For France, infomedfrance@wyeth.com; Trial Manager, Principal Investigator — For Spain, infomed@wyeth.com; Trial Manager, Principal Investigator — For Turkey, Erisc@wyeth.com
Locations (64):
- Australia (3):
  - Nambour, Queensland
  - Cairns
  - Parkville
- Shanghai, China
- Odense, Denmark
- Finland (3):
  - Lahti
  - Seinäjoki
  - Tampere
- France (4):
  - Marseille
  - Nîmes
  - Pierre-Bénite
  - Saint-Denis
- Germany (8):
  - Bochum
  - Frankfurt
  - Freiburg im Breisgau
  - Heidelberg
  - Leipzig
  - Lübeck
  - Münster
  - Tübingen
- Greece (2):
  - Athens
  - Thessaloniki
- Hong Kong (2):
  - New Territories
  - Pokfulam
- India (5):
  - Hyderabad, Telangana
  - Bhopal
  - Lucknow
  - Mumbai
  - New Delhi
- Italy (6):
  - Brescia
  - Genova
  - Pavia
  - Rome
  - Udine
  - Vicenza
- Philippines (2):
  - Manila
  - Quezon City
- Portugal (3):
  - Almada
  - Coimbra
  - Porto
- Riyadh, Saudi Arabia
- South Africa (5):
  - Bellville
  - Kuilsriver
  - Parow
  - Pietermaritzburg
  - Pretoria
- Spain (4):
  - Barcelona
  - Bilbao
  - Madrid
  - Murcia
- Switzerland (4):
  - Bern
  - Geneva
  - Lugano
  - Zurich
- Taiwan (5):
  - Changhua
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District
- Turkey (Türkiye) (2):
  - Ankara
  - Istanbul
- United Kingdom (3):
  - Stockport, Cheshire
  - Birmingham
  - Wigan

REFERENCES:
- [Derived] Qvist N, Warren B, Leister-Tebbe H, Zito ET, Pedersen R, McGovern PC, Babinchak T. Efficacy of tigecycline versus ceftriaxone plus metronidazole for the treatment of complicated intra-abdominal infections: results from a randomized, controlled trial. Surg Infect (Larchmt). 2012 Apr;13(2):102-9. doi: 10.1089/sur.2011.048. Epub 2012 Mar 22. PMID 22439781

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited worldwide from November 2005 to July 2008.
Pre-assignment Details: Patients were screened according to the inclusion/exclusion criteria. Once informed consent was obtained, the patient was enrolled into the study and assigned a randomization number and a treatment regimen.
Groups:
- Tigecycline: Tigecycline administered IV every 12 hours (an initial dose of 100 mg followed by 50 mg every 12 hours).
- Ceftriaxone: Ceftriaxone sodium 2 g administered IV once daily plus metronidazole 1 to 2 g daily in divided IV doses.
Period: Randomization
Arm/Group | Tigecycline | Ceftriaxone
Started | 235 | 238
Completed | 232 | 235
Not Completed | 3 | 3
Not completed — No study drug administered | 3 | 3
Period: Baseline Participants
Arm/Group | Tigecycline | Ceftriaxone
Started | 232 | 235
Completed | 210 | 216
Not Completed | 22 | 19
Not completed — Lost to Follow-up | 5 | 12
Not completed — Death | 6 | 5
Not completed — Withdrawal by Subject | 7 | 1
Not completed — Adverse Event | 1 | 0
Not completed — No bacteria observed | 1 | 0
Not completed — Failure to return | 1 | 1
Not completed — Reintervention | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tigecycline | Ceftriaxone | Total
Number analyzed (Participants) | 232 | 235 | 467
Age Continuous [Mean (Standard Deviation); unit: years] | 48.55 (18.37) | 46.81 (18.38) | 47.67 (18.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 72 | 152
  Male | 152 | 163 | 315

OUTCOME MEASURES:

1. Primary Outcome: Number of Clinically Evaluable (CE) Patients With Clinical Response of Cure at the Test-of-Cure (TOC) Visit
Description: CE population were those who completed TOC assessment of cure or failure (but not indeterminate) or, in case of premature discontinuation due to lack of efficacy, had completed end of treatment assessment such that assessment of clinical response could be made. Clinical response was assigned by investigator per protocol-specified guidelines and defined as: test article and initial intervention (operative and/or radiologically controlled drainage procedure) resolved the intra-abdominal infection. TOC performed 10-28 days after last dose of study drug.
Time Frame: up to 6 weeks
Population: All patients who received at least 1 dose of study drug who had clinical evidence of a complicated intra-abdominal infection (cIAI) and completed the test-of-cure (TOC) assessment of cure or failure within 8 to 44 days after the last administration of study article. Patients with an indeterminate assessment were excluded.
Measure: Number; unit: participants
Arm/Group | Tigecycline | Ceftriaxone
Number analyzed (Participants) | 198 | 189
participants | 162 | 150
Statistical Analysis 1: Comparison: Tigecycline vs Ceftriaxone; Test type: Non-Inferiority or Equivalence — A 2-sided 95% CI (corrected for continuity) was calculated for the true difference between the cure rates. Non-inferiority will be concluded if the lower limit of the 2-sided CI is greater than -15%; t-test, 1 sided; Risk Difference (RD) = 1.6, 95% CI [-6.4 to 9.6] — Estimates of the difference, CI and hypothesis tests are weighted by using minimum risk weights

2. Secondary Outcome: Number of Microbiologically Evaluable (ME) Patients With a Clinical Response of Cure at Test-of-Cure (TOC) Visit
Description: ME population were subjects who were clinically evaluable and had baseline culture with at least 1 identified isolate that was susceptible to study drug and comparator. The clinical response was assigned by the investigator according to the protocol-specified guidelines. A clinical response of cure was defined as: the test article and the initial intervention (operative and/or radiologically controlled drainage procedure) resolved the intra-abdominal infection.
Time Frame: up to 6 weeks
Population: All patients who received ≥1 dose, had clinical evidence of complicated intra-abdominal infection, met all inclusion/exclusion criteria, completed TOC assessment within 8-44 days after last dose, and had a baseline culture with ≥1 identified isolate that was susceptible to both study drugs. Patients with an indeterminate assessment were excluded.
Measure: Number; unit: participants
Arm/Group | Tigecycline | Ceftriaxone
Number analyzed (Participants) | 119 | 108
participants | 97 | 86
Statistical Analysis 1: Comparison: Tigecycline vs Ceftriaxone; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.001, t-test, 1 sided; Risk Difference (RD) = 1.8, 95% CI [-8.8 to 12.5] — Estimates of the difference, CI and hypothesis tests are weighted by using minimum risk weights

3. Secondary Outcome: Number of Microbiologically Evaluable (ME) Patients by Microbiological Response at Test-of-Cure (TOC) Visit
Description: Microbiological response was assessed at patient level was the combined responses for all baseline isolates identified in intra-abdominal and blood cultures. Eradication=baseline isolate not recovered from primary infection site/blood; Presumed Eradication=No sample for culture, clinical response was cure; Persistence=baseline isolate recovered from primary infection site/blood; Presumed Persistence=No sample available for culture, clinical response was failure; Superinfection=culture from primary infection site with new isolate not identified at baseline, clinical response was failure.
Time Frame: up to 6 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Tigecycline | Ceftriaxone
Number analyzed (Participants) | 119 | 108
participants
  Eradication + Presumed Eradication | 98 | 86
  Persistence + Presumed Persistence | 21 | 22
  Superinfection | 3 | 0
Statistical Analysis 1: Comparison: Tigecycline vs Ceftriaxone; Group comparison of eradication + presumed eradication; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; t-test, 1 sided; Risk Difference (RD) = 2.7, 95% CI [-7.9 to 13.3] — Estimates of the difference, CI and hypothesis tests are weighted by using minimum risk weights

4. Secondary Outcome: Number of Days of Inpatient Healthcare Resource Utilization on or Before Test-of-Cure
Description: Healthcare resource utilization assessment included days of overall inpatient hospitalization, days of primary inpatient hospitalization, days of Intensive Care Unit (ICU) treatment and days of non-ICU inpatient hospitalization
Time Frame: up to 6 weeks
Population: All patients who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tigecycline | Ceftriaxone
Number analyzed (Participants) | 232 | 235
days
  Overall inpatient hospitalization | 13.03 (12.45) | 12.69 (10.25)
  Primary inpatient hospitalization | 12.62 (12.28) | 12.16 (9.75)
  ICU treatment | 8.24 (9.47) | 6.14 (8.70)
  Inpatient hospitalization, non-ICU | 11.09 (9.21) | 10.80 (7.93)
Statistical Analysis 1: Comparison: Tigecycline vs Ceftriaxone; Overall inpatient hospitalization; Test type: Superiority or Other; p = 0.750, ANOVA; Treatment as a factor
Statistical Analysis 2: Comparison: Tigecycline vs Ceftriaxone; Primary inpatient hospitalization; Test type: Superiority or Other; p = 0.655, ANOVA; Treatment as a factor
Statistical Analysis 3: Comparison: Tigecycline vs Ceftriaxone; ICU treatment; Test type: Superiority or Other; p = 0.191, ANOVA; Treatment as a factor
Statistical Analysis 4: Comparison: Tigecycline vs Ceftriaxone; Inpatient hospitalization, non-ICU; Test type: Superiority or Other; p = 0.717, ANOVA; Treatment as a factor

ADVERSE EVENTS:
Description: Total # Affected patients includes duplicate patients that had more than one non-serious adverse events.
Arm/Group | Tigecycline | Ceftriaxone
Serious Adverse Events (participants affected / at risk) | 37/232 | 38/235
Other Adverse Events (participants affected / at risk) | 173/232 | 155/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tigecycline (N=232) | Ceftriaxone (N=235)
Infection (General disorders) | 7 | 4
Sepsis (General disorders) | 4 | 5
Abscess (General disorders) | 3 | 3
Septic shock (General disorders) | 4 | 0
Peritonitis (General disorders) | 1 | 2
Abdominal pain (General disorders) | 0 | 2
Fever (General disorders) | 0 | 2
Pain (General disorders) | 0 | 1
Scleroderma (General disorders) | 1 | 0
Traumatic hematoma (General disorders) | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 2
Intestinal perforation (Gastrointestinal disorders) | 1 | 2
Colitis (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 2
Duodenal ulcer hemorrhage (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Blood in stool (Gastrointestinal disorders) | 1 | 0
Cholelithiasis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Intestinal necrosis (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Jaundice (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Liver function tests abnormal (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Healing abnormal (Metabolism and nutrition disorders) | 6 | 5
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Amylase increased (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Pulmonary embolus (Vascular disorders) | 1 | 3
Shock (Vascular disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cerebral ischemia (Vascular disorders) | 1 | 0
Cerebrovascular accident (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Left heart failure (Cardiac disorders) | 0 | 1
Peripheral vascular disease (Vascular disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Acute kidney failure (Renal and urinary disorders) | 1 | 0
Kidney function abnormal (Renal and urinary disorders) | 1 | 0
Urolithiasis (Renal and urinary disorders) | 0 | 1
Local reaction to procedure (Injury, poisoning and procedural complications) | 0 | 2
Disseminated vascular coagulation (Blood and lymphatic system disorders) | 1 | 0
International normalized ratio increased (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tigecycline (N=232) | Ceftriaxone (N=235)
Nausea (Gastrointestinal disorders) | 49 | 50
Vomiting (Gastrointestinal disorders) | 40 | 31
Diarrhea (Gastrointestinal disorders) | 27 | 17
Constipation (Gastrointestinal disorders) | 3 | 8
Infection (General disorders) | 18 | 15
Hypokalemia (Metabolism and nutrition disorders) | 8 | 13
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 8 | 2
Insomina (Nervous system disorders) | 4 | 7
Thrombocythemia (Blood and lymphatic system disorders) | 7 | 6
Local reacation to procedure (Injury, poisoning and procedural complications) | 9 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.